CLINICAL TRIAL: NCT04899089
Title: Cognitive Training in Mild Cognitive Impairment: Effects on Sleep, Cognition and Arousal
Brief Title: Cognitive Training in Mild Cognitive Impairment
Acronym: TRAIN-MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Ashley Curtis, Assistant Professor of Psychiatry, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2053302
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Insomnia; Mild Cognitive Impairment
Keywords: cognitive training; insomnia; mild cognitive impartment; older adults; sleep; cognition
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Video Game Training Condition (Experimental): Participants complete an 8 week long computerized cognitive training intervention. Participants play the games for 45 minutes, three times per week.
  Interventions: Behavioral: Cognitive Training
- Trivia Training Condition (Active Comparator): Participants complete an 8 week long computerized trivia training. Participants complete the trivia training for 45 minutes, three times per week.
  Interventions: Behavioral: Trivia Training

INTERVENTIONS:
Behavioral: Cognitive Training — The computerized training exercises and brain games help stimulate cognitive functions while providing real-time monitoring on the evolution of participants' skills.
  Arms: Video Game Training Condition
Behavioral: Trivia Training — The computerized trivia training asks participants to answer general questions related to pop culture, science, geography, etc. Participants can use online sources to search for answers and will be provided feedback on their accuracy.
  Arms: Trivia Training Condition

SUMMARY:
Older adults (60+ years of age) who meet criteria for mild cognitive impairment and insomnia will be randomly assigned to cognitive training or trivia training and will complete measures of anxiety, sleep, cognition (objective, self-efficacy), and arousal at baseline, and post-intervention. For cognitive training, participants will be provided with login information to access the computerized training, and will complete 8 weeks (45 mins 3x/week) of cognitive training. For trivia training, participants will receive weekly emails that contain trivia assignments that they will complete for 8 weeks (45 mins 3x/week). We will evaluate short-term (i.e., post-training) effects of the two training conditions on subjective anxiety, sleep, arousal, and subjective and objective cognition.

ELIGIBILITY:
Inclusion Criteria:

1. 60+ yrs of age
2. meet criteria for mild cognitive impairment
3. no neurological or psychiatric illness or dementia
4. non-gamers (<2 hour of video/brain training games/week over last 2 yrs)
5. proficient in English (reading and writing)
6. meet clinical dx criteria for Insomnia (e.g., insomnia complaints for 6+ months, complaints occur despite adequate opportunity and circumstances for sleep, consist of one of the following: difficulty falling asleep, staying asleep, or waking up too early, and daytime dysfunction due to insomnia)

Exclusion Criteria:

1. unable to provide informed consent
2. unable to undergo randomization
3. other sleep disorder (e.g., sleep apnea, restless legs syndrome)
4. severe untreated psychiatric comorbidity
5. psychotropic or other medications that alter sleep (unless stabilized for 6 months)
6. uncorrected visual/auditory impairments
7. participation in nonpharmacological tx for sleep/fatigue/mood/cognition outside the current study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Objective Cognition - Computerized Cognitive Tasks | Up to 10 weeks
  Complete computerized tasks. These tasks will measure cognitive functions (e.g., processing speed, attention, memory).
Subjective Cognitive Self-Efficacy. - Cognitive Failures Questionnaire | Up to 10 weeks
  A 25 item questionnaire. Participants rate from 0 (never) to 4 (very often) frequency of cognitive errors. Higher scores indicate lower cognitive self-efficacy.
Subjective Behavioral Sleep- Electronic Daily Sleep Diaries | Up to 10 days
  Electronic Daily Sleep Diaries. Online diaries completed each morning (~5 mins) during the study. Diaries measure sleep onset latency, wake time after sleep onset, total sleep time, and sleep quality.
Subjective Behavioral Sleep- Insomnia Severity Index | Up to 10 weeks
  Brief self-report measure of current perception of insomnia symptom severity, distress and daytime impairment. Commonly used in insomnia treatment outcome research.
Objective Sleep-Watchpat | Up to 10 weeks
  Single night objective sleep recording via a wrist worn device.

SECONDARY OUTCOMES:
Physiological Arousal- Heart Rate Variability | Impact of game related experience will be measured at baseline
  CorSense monitor assessed 5 min heart rate recordings both at rest. Time index variables: SDNN (standard deviation of normal to normal heartbeat intervals)
Anxiety - State-Trait Anxiety Inventory | Up to 10 weeks
  Inventory that asks respondents to rate how true 20 self-descriptive statements (e.g., I feel calm) are on a 4-point scale (1 = not at all, 4 = very much so). Typically, respondents are asked to rate statements according to how they generally feel (trait-anxiety scale) and how they feel in the current moment (state-anxiety scale). Total scores range from 20 to 80, with higher scores indicating greater maladjustment.
Game-related experience- Sessions and duration played | Up to 10 weeks
  During the intervention phase the cognitive training group will play games and will need to log the days and duration played.
Circadian Rhythm- Morningness-Eveningness Questionnaire | Up to 10 weeks
  19-item questionnaire that assesses preference for morning, afternoon, and evening activities. Total score reflects degree of "morningness" or "eveningness" type.
Perceived Stress- Perceived Stress Scale Subjective Arousal- Perceived Stress Scale | Up to 10 weeks
  Perceived Stress Scale is a self-report measure of how life situations are perceived as stressful. The scale consists of 15 items corresponding to everyday situation and participants are asked to rate on a scale from 0 (never) to 4 (very often) how often they felt or thought a specific way. Higher scores correspond to higher perceived stress.
Subjective Arousal- Arousal Predisposition Scale | Up to 10 weeks
  Arousal Predisposition Scale is a 12-item inventory that has been designed to measure the degree to which an individual experiences arousal. Higher scores indicate greater predisposition to arousal.
Game Engagement Questionnaire | Up to 10 weeks
  Questionnaire assessing the experience of the game.
Mood-Depression-Beck Depression Inventory-II | Up to 10 weeks
  21-item inventory that asks respondents to rate on a scale of 0 (no depressive feelings) to 3 (most depressive feelings) their feelings towards various aspects of daily living/situations. Higher total scores indicate worse depressive symptoms.
Alcohol Use - Alcohol Use Disorder Test | Baseline
  10-item questionnaire that assess the frequency of alcohol use and problems associated with alcohol use over the past year.
Physical Activity - International Physical Activity Questionnaire | Up to 10 weeks
  7- item questionnaire assessing the different kinds of physical activities that the participant does as pat of their everyday life.
Personality - Big Five Inventory | Baseline
  10 question assessment measuring personality
Computer Proficiency- Computer Proficiency Questionnaire | Baseline
  This questionnaire asks about participants' ability to perform a number of tasks with a computer. Will be examined as a covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Curtis, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be assigned a participant number and de-identified. De-identified data will be shared with other researchers.